CLINICAL TRIAL: NCT00003184
Title: Phase I Trial Using a CD80-Modified Allogeneic Breast Cancer Cell Line to Vaccinate HLA-A2-Positive Women With Breast Cancer
Brief Title: Vaccine Therapy in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066010; PPMC-IRB-94-78; OCC-ONC-9408-L; NCI-V98-1379
Record Dates: First submitted 1999-11-01; First posted 2003-07-11 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2000-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BCG Vaccine; sargramostim

INTERVENTIONS:
Biological: BCG vaccine
Biological: CD80 breast cancer vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines made from breast cancer cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccines made from breast cancer cells in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of vaccination strategies employing a CD80-transfected allogeneic breast cancer cell line (MDA-MB-231).
* Assess the immunologic response of lymphocytes isolated from lymph nodes draining the vaccination site following a single dose of CD80-transfected MDA-MB-231.
* Assess the development of systemic immunity following multiple injections of CD80-transfected MDA-MB-231.
* Observe for tumor regression.

OUTLINE: This is a dose-escalation study.

Patients receive intradermal vaccinations containing CD80-transfected cells with or without sargramostim (GM-CSF) or with or without BCG. Vaccinations are administered every 2 weeks for 6 weeks and then monthly for 3 months. Patients may receive 1 of 2 different doses of GM-CSF. GM-CSF is administered with the vaccination, then every 12 hours for 7 days. Monthly vaccinations may continue as long as response is shown.

Cohorts of 5 patients each are treated at each dose/combination. Each cohort completes treatment before the next cohort is accrued.

Patients are followed at weeks 4 and 8, then every 2 months for 6 months, then every 3 months for 1 year, and then every 6 months until disease progression.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic breast cancer

  * Stage IV disease patients who have either been treated to maximal response or who have had high dose chemotherapy or a marrow ablative regimen (if they meet immunologic criteria and have not received more than 2 chemotherapy regimens for treatment of metastatic disease)
  * Patients with advanced stage disease who:

    * Received at least 1 standard chemotherapy regimen, but no more than 2, for treatment of metastatic disease
    * Refused chemotherapy
    * Refused or progressed despite hormonal therapy
* Measurable or evaluable disease
* Positive or negative for HLA-A2
* Must have superficial inguinal or axillary lymph nodes that are free of tumor involvement and are surgically accessible
* No symptomatic or acutely life threatening tumor that is judged likely to require intervention with alternative modalities within 3 months
* No brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3

Hepatic:

* Not specified

Renal:

* BUN less than 25 mg/dL
* Creatinine less than 1.8 mg/dL

Cardiovascular:

* No ischemic or congestive cardiac disease requiring chronic medication
* No New York Heart Association class III or IV heart disease
* No evidence of ischemic change or ventricular ectopy (greater than 4/min) on electrocardiogram (EKG)
* No evidence of type II arterial-ventricular block
* No evidence of current cardiac disease by stress test and EKG

Other:

* HIV negative
* No active infection requiring treatment
* No psychiatric illness
* No history of seizure disorder
* No other prior malignancy within the past 10 years except squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior specific or nonspecific immunotherapy, unless there is obvious progression of metastatic disease, and recovered

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy, unless there is obvious progression of metastatic disease, and recovered

Endocrine therapy:

* At least 4 weeks since prior steroids, unless there is obvious progression of metastatic disease, and recovered

Radiotherapy:

* Concurrent radiotherapy allowed for local control of disease

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-08; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Urba, MD, PhD, Study Chair — Providence Cancer Center, Earle A. Chiles Research Institute
Locations (1):
- Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon, United States

REFERENCES:
- [Result] Schoof DD, Smith JW 2nd, Disis ML, Brant-Zawadski P, Wood W, Doran T, Johnson E, Urba WJ. Immunization of metastatic breast cancer patients with CD80-modified breast cancer cells and GM-CSF. Adv Exp Med Biol. 1998;451:511-8. doi: 10.1007/978-1-4615-5357-1_79. No abstract available. PMID 10026920